CLINICAL TRIAL: NCT00106106
Title: Acamprosate for Central Nervous System Hyperexcitability and Neuroadaptation in Alcohol Withdrawal
Brief Title: Acamprosate to Reduce Symptoms of Alcohol Withdrawal
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Markus Heilig, Clinical Director, National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 050120; 05-AA-0120 (Other: National Institutes of Health)
Record Dates: First submitted 2005-03-19; First posted 2005-03-21 (Estimated); Results first posted 2012-01-05 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2012-01

CONDITIONS: Alcohol-Related Disorders; Alcohol Dependence; Alcoholism; Healthy Volunteer
Keywords: Alcoholism; Acamprosate; Withdrawal; Glutamate; Magnetic Resonance Spectroscopy; Alcohol Dependence; Healthy Volunteer; HV
MeSH Terms: conditions — Alcohol-Related Disorders; Alcoholism | interventions — Magnetic Resonance Spectroscopy; Acamprosate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): For subjects randomized to placebo control, placebo doses were given every 8 hours.
  Interventions: Procedure: NMR-spectroscopy
- Acamprosate (Experimental): For subjects randomized to active treatment, the first 3 acamprosate doses were 1332 mg every 8 hours in an attempt to more rapidly achieve active plasma concentrations, followed by 666 mg acamprosate every 8 hours for the remainder of the study.
  Interventions: Procedure: NMR-spectroscopy; Drug: Oral acamprosate

INTERVENTIONS:
Procedure: NMR-spectroscopy — Scans were performed on a 3T scanner using the echo-time-averaged PRESS sequence previously published to detect glutamate's resonance line at 2.35 ppm and average out the interferences from glutamine, NAA and the macromolecules.
  Other Names: Magnetic Resonance Spectroscopy; MRS
Drug: Oral acamprosate — For subjects randomized to active treatment, the first 3 acamprosate doses were 1332 mg every 8 hours in an attempt to more rapidly achieve active plasma concentrations, followed by 666 mg acamprosate every 8 hours for the remainder of the study.
  Other Names: Campral
  Arms: Acamprosate

SUMMARY:
This study will examine whether a new drug called acamprosate can be helpful for alcohol withdrawal, a result of drinking high amounts of alcohol for long periods of time. Alcohol withdrawal can cause various symptoms, including nausea or vomiting, anxiety or depression, tremor, high blood pressure, and others. During withdrawal, brain chemicals called neurotransmitters change, with some rising to abnormally high levels. These changes may contribute to alcohol craving, drinking relapse and impaired mental performance. This study will see if taking acamprosate for 4 weeks can lower the levels of neurotransmitters, such as glutamate, lessen withdrawal symptoms and decrease alcohol craving and brain damage associated with withdrawal.

Healthy normal volunteers and alcohol-dependent patients between 21 and 65 years of age may be eligible for this study.

Participants are admitted to the hospital for 28 days. They receive standard inpatient care for alcohol detoxification, including a medical history and physical examination, neurological evaluation, laboratory tests, nursing, nutrition, discharge planning and referrals for treatment of concomitant conditions, if needed. In addition, they are randomly assigned to take either two acamprosate or two placebo pills three times a day for 28 days and undergo the following tests and procedures:

* Days 1-28: Drug treatment. Patients take acamprosate or placebo daily. Patients with severe withdrawal symptoms may also receive diazepam (Valium). Throughout their hospitalization, patients fill out questionnaires about their emotional state and personality and are interviewed by staff about their mental health, use of alcohol, cigarettes, and illicit drugs, employment, support systems and family and social relationships, and their legal status.
* Days 2 and 3: Blood tests. Blood is tested for levels of the stress hormones cortisol and ACTH, which are released to excess during alcohol withdrawal. For this test, a heparin lock (thin, flexible plastic tube with a rubber stopper on the end) is placed in an arm vein for blood collections each day at 6 AM, 12 noon, 6 PM and 12 midnight. Patients rest in bed for 30 minutes before each collection.
* Day 4: Magnetic resonance imaging (MRI) and magnetic resonance spectroscopy (MRS). These procedures are done at the same time. They use a strong magnetic field and radio waves to show structural and chemical changes in the brain. The patient lies on a table in a space enclosed by a metal cylinder (the scanner) for about 20 to 30 minutes during the test.
* Day 5: Lumbar puncture (spinal tap). A local anesthetic is given to numb the area for the procedure. Then, a needle is inserted in the space between the bones in the lower back where the cerebrospinal fluid circulates below the spinal cord. A small amount of fluid is collected through the needle.
* Days 5 and 6: Dexamethasone-corticotropin releasing factor (CRF) test. This test measures the effect of alcohol withdrawal on ACTH and cortisol. The patient takes a standard dose of the steroid dexamethasone at 11 PM on day 5. At noon the next day, they are given lunch and then stay in bed and rest. A plastic tube is put in an arm vein. A salt water solution is slowly infused through the catheter and a blood sample is withdrawn through it. At 3 p.m., the patient is given 100 micrograms of the hormone CRF. Repeated blood samples are obtained to measure ACTH and cortisol.
* Days 23-27: All of the tests done on days 2-6 are repeated, except the MRI. MRS is repeated to measure neurotransmitters.

DETAILED DESCRIPTION:
Objective: Clinical as well as preclinical studies indicate that the process of developing alcohol dependence recruits a progressively aggravated hyperglutamatergic state, which in turn is a key signal for emotional dysregulations leading to craving and relapse, as well as neurotoxicity leading to cognitive impairment and loss of grey matter in alcoholic patients. Acamprosate has recently been approved for relapse prevention in sober alcoholics, an effect mediated through largely unknown mechanisms. Preclinical data indicate, however, that it might primarily be useful for targeting the hyperglutamatergic state that develops during recurring withdrawal episodes, halting the process described above. If so, acamprosate might be of value as a withdrawal treatment to prevent the progression of alcohol dependence. The aim of the present protocol is to evaluate, in a randomized controlled trial, the effects of acamprosate during withdrawal and the early post-withdrawal phase. The primary outcome variable will be central glutamate/glutamine concentration as determined by MR spectroscopy. A number of exploratory biological and clinical measures will in addition be obtained and used for secondary analyses as specified below.

Study Population: We will study patients age 21 - 65, without gross impairment of judgment or complicated psychiatric or other morbidity, going into withdrawal or with a high probability of doing so, will be admitted as inpatients to the NIAAA CC-unit. A group of healthy volunteers who do not receive study medication will be examined separately in order to confirm that a hyperglutamatergic state is present in the patients during withdrawal.

Design: All patients will receive standard care for alcohol detoxification. In addition, half of them will be randomized in a blinded fashion to oral acamprosate, two 333 mg tablets taken 3 times daily or corresponding placebo. Validated rating scales (CIWA-Ar, CPRS-SA) will be used to assess intensity of withdrawal and psychopathology. If severity of withdrawal exceeds a predefined criterion, standard diazepam treatment will be added to study medication. The accrual target is based on a primary analysis sample of patients who will not require diazepam medication, which is a potential confound. A secondary analysis will be carried out on the complete sample, analyzing the requirement for/amount of diazepam supplement as a secondary outcome variable.

Outcome Measures: A battery of tests will be obtained during the 1st and 3rd week of inpatient treatment. These will include NMR-spectroscopy to quantify central levels of excitatory and inhibitory amino acids (primary outcome variable: GluX concentration); lumbar puncture to obtain CSF for analysis of neurotransmitter/neurohormone metabolites and synaptic proteins. Repeated 4 x daily blood collection for analysis of serum cortisol and ACTH will be obtained to assess spontaneous activity and circadian variation of the HPA-axis, and the combined dexamethasone - CRH test will be carried out to dynamically probe this system, and gauge its sensitivity for feedback inhibition.

ELIGIBILITY:
* INCLUSION CRITERIA - PATIENTS:

  1. Alcohol dependence according to DSM-IV, based on the alcohol dependence module of the SCID I-interview, and alcohol withdrawal, based on either of:

     Clinically manifest significant alcohol withdrawal symptoms, with or without detectable blood alcohol concentrations.

     In absence of the above, current intoxication above 0.1 g/dl BAC, self-reported history of continuous alcohol use > 1 month, and self-reported previous episodes of significantly distressful alcohol withdrawal symptoms, whether treated or not.
  2. Age 21 - 65; in younger subjects, maturation processes of the central nervous system are still ongoing; while in older subjects, degenerative changes may confound the measures studied.
  3. Smoking status: this will be noted and evaluated using the Fagerstrom inventory, so that its potential contribution to group differences can be assessed. This variable will not otherwise affect inclusion / exclusion.

INCLUSION CRITERIA - HEALTHY CONTROLS:

Subjects will be eligible for inclusion if they are aged 21-65. They will be as closely as possible matched to the patient population with regard to gender and age.

EXCLUSION CRITERIA - PATIENTS:

1. Current or prior history of any disease, including cardiovascular, respiratory, gastrointestinal, hepatic, renal, endocrine, or reproductive disorders, or a positive hepatitis or HIV test at screening.
2. Current Axis-I psychiatric illness.
3. Current or prior history of any alcohol or drug dependence, as well as non-drinkers (alcohol-naive individuals or current abstainers).
4. Positive result on urine screen for illicit drugs.
5. Nursing, pregnancy or intention to become pregnant for women. Female participants will undergo a urine beta-hCG test to ensure they are not pregnant.
6. Pregnancy (negative test required) or ongoing breastfeeding.
7. Use of prescription or OTC medications know to interact with alcohol within 2 weeks of the study. These include, but may not be limited to: isosorbide, nitroglycerine, benzodiazepines, warfarin, anti-depressants such as amitriptyline, clomipramine and nefazodone, anti-diabetes medications such as glyburide, metformin and tolbutamide, H2-antagonists for heartburn such as cimetidine and ranitidine, muscle relaxants, anti-epileptics including phenytoin and Phenobarbital codeine, and narcotics including darvocet, percocet and hydrocodone. Drugs known to inhibit or induce enzymes that metabolize alcohol should not be used for 4 weeks prior to the study. These include chlorzoxazone, isoniazid, metronidazole and disulfiram. Cough-and-cold preparations which contain anti-histamines, pain medicines and anti-inflammatories such as aspirin, ibuprofen, acetaminophen, celecoxib and naproxen, should be withheld for at least a 72 hours prior to each study session.
8. Self-reported history of flushing upon intake of alcohol.
9. Inability to undergo an MR scan, due to presence of ferromagnetic objects in their bodies which could cause adverse effects in the MRI scanner, pronounced anxiety provoked by enclosed spaces, or other reasons.

EXCLUSION CRITERIA - HEALTHY CONTROLS:

1. History of any substance use disorder.
2. Average weekly consumption over last 4 weeks, assessed with Time-Line Follow-Back, exceeding 210g pure alcohol / week, or consumption of more than 60g pure alcohol on any single occasion within last 3 days
3. Any history of a psychotic disorder or a history of any other psychiatric diagnosis within the last 12 months
4. Any prescription medication within the last 2 months
5. Pregnant (negative pregnancy test required) or breastfeeding
6. Inability to undergo an MR scan, due to presence of ferromagnetic objects in their bodies which could cause adverse effects in the MRI scanner, pronounced anxiety provoked by enclosed spaces, or other reason

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2005-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Daeppen JB, Gache P, Landry U, Sekera E, Schweizer V, Gloor S, Yersin B. Symptom-triggered vs fixed-schedule doses of benzodiazepine for alcohol withdrawal: a randomized treatment trial. Arch Intern Med. 2002 May 27;162(10):1117-21. doi: 10.1001/archinte.162.10.1117. PMID 12020181
- [Background] Liskow BI, Goodwin DW. Pharmacological treatment of alcohol intoxication, withdrawal and dependence: a critical review. J Stud Alcohol. 1987 Jul;48(4):356-70. doi: 10.15288/jsa.1987.48.356. PMID 2956463
- [Background] Mayo-Smith MF. Pharmacological management of alcohol withdrawal. A meta-analysis and evidence-based practice guideline. American Society of Addiction Medicine Working Group on Pharmacological Management of Alcohol Withdrawal. JAMA. 1997 Jul 9;278(2):144-51. doi: 10.1001/jama.278.2.144. PMID 9214531
- [Derived] Vatsalya V, Cave MC, Kumar R, Srivastava S, Khanal S, Jenson AB, Schwandt ML, Barve SS, Ramchandani VA, McClain CJ. Alterations in Serum Zinc and Polyunsaturated Fatty Acid Concentrations in Treatment-Naive HIV-Diagnosed Alcohol-Dependent Subjects with Liver Injury. AIDS Res Hum Retroviruses. 2019 Jan;35(1):92-99. doi: 10.1089/AID.2018.0124. Epub 2018 Dec 11. PMID 30280905
- [Derived] Vatsalya V, Kong M, Cave MC, Liu N, Schwandt ML, George DT, Ramchandani VA, McClain CJ. Association of serum zinc with markers of liver injury in very heavy drinking alcohol-dependent patients. J Nutr Biochem. 2018 Sep;59:49-55. doi: 10.1016/j.jnutbio.2018.05.003. Epub 2018 May 12. PMID 29960116
- [Derived] Umhau JC, Momenan R, Schwandt ML, Singley E, Lifshitz M, Doty L, Adams LJ, Vengeliene V, Spanagel R, Zhang Y, Shen J, George DT, Hommer D, Heilig M. Effect of acamprosate on magnetic resonance spectroscopy measures of central glutamate in detoxified alcohol-dependent individuals: a randomized controlled experimental medicine study. Arch Gen Psychiatry. 2010 Oct;67(10):1069-77. doi: 10.1001/archgenpsychiatry.2010.125. PMID 20921123

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Acamprosate
Started | 26 | 23
Completed Both MRS Scans | 18 | 15
Completed | 22 (Although 22 subjects completed all other assessments for the study, only 18 completed both MRS scans) | 19 (Although 19 subjects completed all other assessments for the study, only 15 completed both MRS scans)
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Acamprosate | Total
Number analyzed (Participants) | 26 | 23 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 23 | 49
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 35.1 (6.1) | 35.0 (5.8) | 35.1 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 15 | 15 | 30
Region of Enrollment [Number; unit: participants]
  United States | 26 | 23 | 49

OUTCOME MEASURES:

1. Primary Outcome: Ratio of Glutamate to Creatine in the Anterior Cingulate of the Brain, Measured on Day 4
Description: The ratio of glutamate to creatine was determined using magnetic resonance spectroscopy (MRS), a technique that complements magnetic resonance imaging (MRI). MRS is used to determine the concentration of brain metabolites, such as glutamate, in brain tissue. MRS utilizes a magnetic field to look at magnetic nuclei, which absorb and re-emit electromagnetic energy in the presence of the magnetic field. By looking at the peaks in the resultant spectra the structure and concentration of metabolites can be determined.
Time Frame: Day 4
Population: The analysis of participants was per protocol, i.e., all subjects who completed two MRS scans(Day 4 and Day 25) and for whom there were two measures of the glutamate/creatine ratio
Measure: Mean (Standard Error); unit: Ratio of glutamate to creatine
Arm/Group | Placebo | Acamprosate
Number analyzed (Participants) | 18 | 15
Ratio of glutamate to creatine | 1.256772 (0.038924) | 1.294178 (0.043249)

2. Primary Outcome: Ratio of Glutamate to Creatine in the Anterior Cingulate of the Brain, Measured on Day 25
Description: as for outcome 1
Time Frame: Day 25
Measure: Mean (Standard Error); unit: Ratio of glutamate to creatine
Arm/Group | Placebo | Acamprosate
Number analyzed (Participants) | 18 | 15
Ratio of glutamate to creatine | 1.350375 (0.044497) | 1.166667 (0.049441)

ADVERSE EVENTS:
Arm/Group | Placebo | Acamprosate
Serious Adverse Events (participants affected / at risk) | 0/26 | 1/23
Other Adverse Events (participants affected / at risk) | 20/22 | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=26) | Acamprosate (N=23)
Vaso-vagal faint (General disorders) | 0 (0) | 1 (1) — Following an uneventful lumbar puncture and a brief smoking break, the female patient felt faint when she sat down to eat. A nurse had her lie down on the floor until she recovered.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=22) | Acamprosate (N=19)
Abnormal Dreaming (Nervous system disorders) | 11 | 11
Anxiety (Nervous system disorders) | 9 | 12
Decreased interest in sex (Nervous system disorders) | 6 | 6
Diarrhea (Gastrointestinal disorders) | 3 | 6
Dizziness (Nervous system disorders) | 5 | 6
Feeling Down (Nervous system disorders) | 9 | 11
Headaches (General disorders) | 7 | 12
Impaired concentration (Nervous system disorders) | 7 | 7
Lack of appetite (Gastrointestinal disorders) | 3 | 7
Lack of energy (General disorders) | 7 | 10
Mood swings (Nervous system disorders) | 9 | 13
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 3
Nausea (Gastrointestinal disorders) | 2 | 3
Nervousness (Nervous system disorders) | 7 | 10
Sensation of prickling or tingling on the skin (Nervous system disorders) | 6 | 2
Shakiness (Nervous system disorders) | 3 | 7
Sleepiness (Nervous system disorders) | 15 | 13
Sleeplessness (Nervous system disorders) | 10 | 12
Stomach aches (General disorders) | 2 | 8
Vomiting (Gastrointestinal disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No